CLINICAL TRIAL: NCT01043328
Title: Comparison of Detection of Human Papillomavirus on Tissue, Saliva and Serum
Brief Title: Human Papillomavirus on Oral Tissue, Saliva and Serum
Acronym: CDHPOTSS
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Principal Investigator, Adriana Demathé, PhD Adriana Demathe, UPECLIN HC FM Botucatu Unesp
Other Study IDs: upeclin/FOA-Unesp-05
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Squamous Cell Carcinoma
Keywords: human papillomavirus; nested PCR; saliva; serum; oral tissues
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — This biospecimens will be retained: whole blood, exfoliated cells, saliva and formalin-fixed paraffin-embedded tissues.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GROUP OSCC: The study group is composed by patients with a condition that requires a procedure/surgery for oral squamous cell carcinoma treatment.
  INTERVENTIONS: Collect blood, saliva and oral tissue.
- CONTROL GROUP: Group without oral squamous cell carcinoma but with a condition that requires prosthetic procedure/surgery.
  INTERVENTIONS: Collect blood, saliva and oral tissue.

SUMMARY:
Human papillomavirus (HPV) is one of the most prevalent infections in the world with several millions of new cases diagnosed yearly. Oral HPV infection may be associated with different diseases of oral cavities including some cases of oropharyngeal cancer.

The aim of this report is to detect the presence of HPV DNA in samples of biopsies, oral swabs, saliva and serum of patient with oral squamous cell carcinoma (OSCC) and controls. We hoped to find there is correlation among the presence of HPV DNA in the several biological materials and if it is possible to use the saliva as screening to HPV DNA detection. The presence of tumor HPV DNA in blood may be of diagnostic and prognostic value.

DETAILED DESCRIPTION:
This study will made at the buccal cancer center of UNESP and involved forty patients (n = 40) and forty controls. Serum samples, oral swabs and saliva will collect at the date of diagnosis before therapy and will store at -80 ºC until analysis. Formalin-fixed paraffin-embedded oral squamous cell carcinoma tissues and other biologic samples will process with phenol/chloroform extraction method.

Tumors from 40 OSCC patients at the UNESP University will be obtained from biopsy with prior consent, along with corresponding venipuncture blood, saliva collection and exfoliated buccal cells samples. From controls will be obtained all samples except biopsy tissues. Clinical information including tumor location, stage, and nodal status will be recorded.

Clotted blood specimens will be centrifuged at low speed for 5 min, and the serum was stored at - 80 °C before DNA extraction. Serum samples (400 ml) will be used for DNA extraction. Whole saliva and exfoliated buccal cells will be digested in proteinase K at 48°C during two hours, serum and tumor tissue samples will be digested in proteinase K at 48°C overnight, followed by phenol/chloroform extraction and ethanol precipitation of DNA for all samples. After resuspension in 50 ml of distilled water, the mean working DNA concentrations will be 100-150 ng/ml per serum and tissues samples and 30-50 ng/ ml per whole saliva and exfoliated buccal cells samples. For beta-globin PCR will be used 150 to 300 ng of purified total cellular DNA, to assess the quality of the DNA using the PCR primers GH20 and PC04. After confirmation of the presence and integrity of genomic human DNA, the same amount of DNA will be testing for HPV DNA by nested polymerase chain reaction (PCR) in all samples. In first PCR round degenerate consensus primers MY11 and MY09 will be using to amplify fragments of 450 bp. HPV DNA will amplified in a second round by GP5+ and GP6+ primer sets. The other reaction components will be: 10.9 microlitres of ultra-pure water, 2.5 microlitres PCR buffer 10X, 4mM MgCl2, 15 pmol dNTPs and 1 unit of Platinum Taq DNA polymerase. Approximately 150-300 ng of genomic DNA from each sample will be add to the mixture. The same amount of Hela cells, with up to 4 copies of HPV-18 per cell, will be used as positive control for HPV infection. The negative control will be composed by all PCR components except DNA. The mixture underwent initial denaturation to 94ºC for 10 min, before 40 PCR cycles (94ºC for 1 min; 55ºC for 1 min; 72ºC for 40) and 72°C for 4 minutes. For nPCR, two microliters of the product from the first reaction will be used directly in a reaction containing: 0,02 mM of each primer GP5+ and GP6+(Invitrogen Life Technologies®, Brazil), which produce a 150 pb DNA fragment. The remaining reaction components and conditions will be as described for the first round of PCR, except for the annealing temperature that will be reduced to 43ºC. Ten microliters of the nPCR products will be fractionated by electrophoresis in a 8% polyacrylamide gel, for 3 hours at 100 volts. Band visualization will be performed by staining with silver nitrate solution. Samples will be scored as either HPV DNA-positive or negative based on the inspection of silver nitrate stained bands. PCR amplification will be performed in triplicates for each sample. Samples will be classified as positive or negative based on gel analysis.

Differences in proportion will be evaluated by means of Fisher's exact test. A P value of less then 0.05 will be considered statistically significant. These statistical calculations will be performed using SPSS, version 10.0, for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of squamous cell carcinoma, presented lesions with primary site in the mouth or oropharynx;
* Matched controls without a condition.

Exclusion Criteria:

* Patients that received radiotherapy.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: university dental care clinic patients with or without a condition
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
DNA HPV status (positive/negative) | six months

SECONDARY OUTCOMES:
clinical and pathological characteristics | six months

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Demathe, PhD, Principal Investigator — UNESP Dental School; Glauco I Miyahara, PhD, Study Director — UNESP Dental School
Locations (1):
- Glauco Issamu Miyahara, Araçatuba, São Paulo, Brazil

REFERENCES:
- [Background] Bodaghi S, Wood LV, Roby G, Ryder C, Steinberg SM, Zheng ZM. Could human papillomaviruses be spread through blood? J Clin Microbiol. 2005 Nov;43(11):5428-34. doi: 10.1128/JCM.43.11.5428-5434.2005. PMID 16272465
- [Background] Zhao M, Rosenbaum E, Carvalho AL, Koch W, Jiang W, Sidransky D, Califano J. Feasibility of quantitative PCR-based saliva rinse screening of HPV for head and neck cancer. Int J Cancer. 2005 Nov 20;117(4):605-10. doi: 10.1002/ijc.21216. PMID 15929076